CLINICAL TRIAL: NCT02230371
Title: The Serotonin Receptor Type 3 Antagonist Granisetron as a New Treatment Approach for Patients With Chronic Myofascial Pain in the Orofacial Muscles
Brief Title: Study on the Effect of Granisetron on Myofascial Pain in the Orofacial Muscles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Folktandvården Stockholms län AB (Other Government)
Responsible Party: Principal Investigator, Nikolaos Christidis, Assistant professor, PhD, DDS, Senior Consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NC3; 2005-006042-41 (EudraCT Number)
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Myofascial Pain; Temporomandibular Disorders
Keywords: Myofascial pain; TMD; 5-HT3; Granisetron; Placebo-controlled; Patients; Randomized; Double-blind
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Granisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Granisetron (Experimental): Granisetron (Kytril®; 1 mg/mL, Roche, Stockholm, Sweden) is injected into a maximum of six muscle sites in each patient. The most painful sites to palpation of the masticatory muscles is chosen, either in the same muscle (maximum 3 sites per muscle) or in a different. The injected volume into each site is0.5 mL, hence the maximum dose of granisetron a patient can receive is 3 mg per treatment. This is repeated after one and two weeks.
  Interventions: Drug: Granisetron
- Control (placebo) (Placebo Comparator): Placebo (isotonic saline (NaCl); 0.9 mg/mL, Fresenius Kabi, Uppsala, Sweden) is injected into a maximum of six muscle sites in each patient. The most painful sites to palpation of the masticatory muscles is chosen, either in the same muscle (maximum 3 sites per muscle) or in a different. The injected volume into each site is 0.5 mL. This is repeated after one and two weeks.
  Interventions: Drug: Control (placebo)

INTERVENTIONS:
Drug: Granisetron — If the patient does not have any pain after the first or second injection of granisetron (Kytril®; 1 mg/mL, Roche, Stockholm, Sweden), there will be no more injections but the patient will still come for the follow ups.
  Other Names: Kytril (Roche)
  Arms: Granisetron
Drug: Control (placebo) — If the patient does not have any pain after the first or second injection of granisetron (isotonic saline (NaCl); 0.9 mg/mL, Fresenius Kabi, Uppsala, Sweden), there will be no more injections but the patient will still come for the follow ups.
  Other Names: Isotonic saline 9%
  Arms: Control (placebo)

SUMMARY:
The aim of this study is to to investigate if local treatment with intramuscular injections of granisetron are effective in alleviating pain in patients with chronic myofascial pain in the orofacial muscles

The study hypothesis is that local administration of granisetron reduces pain and allodynia/hyperalgesia in patients with chronic myofascial pain in the orofacial muscles and that this effect of granisetron on pain is larger than the effect from placebo

DETAILED DESCRIPTION:
This randomized, placebo-controlled, double blind trial (RCT) is carried out during the period of May 2006 to December 2014 as a multicenter study. The two participating centers are the Section of Orofacial Pain and Jaw Function, Department of Dental Medicine, Karolinska Institutet, Sweden and Department of Clinical Oral Physiology at the Eastman Institute, Folktandvården Stockholms län AB, Stockholm, Sweden. The patients are divided randomly into two groups that receive either granisetron or placebo. The randomization is performed by computer (www.randomization.com) by a research assistant not participating in data collection.

The study comprise seven visits; V1) Screening for study participation, V2) First treatment, V3) Second treatment, V4) Third treatment, and V5 to V7) Follow-ups at 1, 2 and 12 months (Fig. Y1) V1 (baseline) include a general health questionnaire, the RDC/TMD Axis II questionnaires (25), the McGill Pain Questionnaire (MPQ) (27), pain drawings of the lateral side of the head (each side separately), and a 1-week pain diary. In addition, a clinical examination according to the RDC/TMD Axis I is performed, including registration of the maximum voluntary mouth opening capacity (MUMO), and also registration of the pressure pain threshold (PPT) as well as blood sampling.

V2-V4 include a shortened clinical examination according to RDC including registration of MUMO and PPT, treatment with intramuscular injections of study substance and a 1-week pain diary. At V3 and V4 a patient's global assessment of treatment outcome questionnaire is also included.

V5-V7 include the RDC/TMD Axis II questionnaires, the McGill Pain Questionnaire (MPQ), pain drawings of the lateral side of the head (each side separately), a 1-week pain diary, a patient's global assessment of treatment outcome questionnaire, a clinical examination according to the RDC/TMD Axis I including registration of MUMO and PPT, and registration of adverse events.

Three orofacial pain specialists (N.C., L.F., B.H.M.) and one dentist attending a specialist training program (S.O.) will be calibrated in the RDC/TMD examination technique to a gold standard examiner (M.E.) during one day, and will perform the study. They and the patients are blinded to group assignment (i.e. study substance) during the entire trial and the substances used will not be revealed until the last patient has undergone the last follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* a diagnosis of myofascial pain according to the research diagnostic criteria for TMD Axis I (RDC/TMD)
* duration of TMD pain ≥ 3 months
* self-assessed average myofascial-TMD pain intensity of ≥ 30 mm on a 100-mm visual analogue scale (VAS) during one week prior to examination
* familiar pain upon digital palpation of the masseter and/or the temporalis muscles.
* The patients remain included with one or several co-diagnoses of; a) disc displacement with or without reduction, b) osteoarthrosis in the any of the temporomandibular joints (TMJ), and c) episodic or chronic tension type headache

Exclusion Criteria:

* diagnosed systemic muscular or joint diseases (e.g. fibromyalgia, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis)
* whiplash associated disorder
* neuropathic pain or neurological disorders (e.g. myasthenia gravis, orofacial dystonia)
* history of psychiatric disorders
* pain of dental origin
* use of muscle relaxants or any medication that might influence the response to pain
* pregnancy or lactation
* known hypersensitivity to granisetron

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks after treatment
  Change of the median weekly pain intensity compared to baseline A 100-mm VAS is used for each day of the week
Pain intensity | 6 months after treatment
  Change of the median weekly pain intensity compared to baseline A 100-mm VAS is used for each day of the week

SECONDARY OUTCOMES:
Physical and emotional functioning | 8 weeks after treatment
  Assessed with Axis II of the RDC/TMD (research diagnostic criteria for temporomandibular disorders), including the questionnaires:
  Graded Chronic Pain Scale SCL-90R
Physical and emotional functioning | 6 months after treatment
  Assessed with Axis II of the RDC/TMD (research diagnostic criteria for temporomandibular disorders), including the questionnaires:
  Graded Chronic Pain Scale SCL-90R
Adverse events | 1 week after the first injection
  Any possible adverse event is registered
Adverse events | 1 week after the second injection
  Any possible adverse event is registered
Adverse events | 1 week after the third injection
  Any possible adverse event is registered
Adverse events | 8 weeks after the third injection
  Any possible adverse event is registered
Adverse events | 6 months after the third injection
  Any possible adverse event is registered

OTHER OUTCOMES:
Changes in pressure pain threshold | 8 weeks after treatment
  Assessed with a digital algometer (Somedic Sales, Hörby, Sweden)
Changes in pressure pain threshold | 6 months after treatment
  Assessed with a digital algometer (Somedic Sales, Hörby, Sweden)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Christidis, PhD, DDS, Principal Investigator — Karolinska Institutet, Department of Dental Medicine
Locations (1):
- Karolinska Institutet, Department of Dental Medicine, Huddinge, Sweden

REFERENCES:
- [Background] Christidis N, Kopp S, Ernberg M. The effect on mechanical pain threshold over human muscles by oral administration of granisetron and diclofenac-sodium. Pain. 2005 Feb;113(3):265-270. doi: 10.1016/j.pain.2004.10.016. PMID 15661432
- [Background] Christidis N, Nilsson A, Kopp S, Ernberg M. Intramuscular injection of granisetron into the masseter muscle increases the pressure pain threshold in healthy participants and patients with localized myalgia. Clin J Pain. 2007 Jul-Aug;23(6):467-72. doi: 10.1097/AJP.0b013e318058abb1. PMID 17575485
- [Background] Ernberg M, Lundeberg T, Kopp S. Effect of propranolol and granisetron on experimentally induced pain and allodynia/hyperalgesia by intramuscular injection of serotonin into the human masseter muscle. Pain. 2000 Feb;84(2-3):339-46. doi: 10.1016/s0304-3959(99)00221-3. PMID 10666539
- [Background] Ernberg M, Lundeberg T, Kopp S. Pain and allodynia/hyperalgesia induced by intramuscular injection of serotonin in patients with fibromyalgia and healthy individuals. Pain. 2000 Mar;85(1-2):31-9. doi: 10.1016/s0304-3959(99)00233-x. PMID 10692600
- [Background] Ernberg M, Hedenberg-Magnusson B, Alstergren P, Kopp S. The level of serotonin in the superficial masseter muscle in relation to local pain and allodynia. Life Sci. 1999;65(3):313-25. doi: 10.1016/s0024-3205(99)00250-7. PMID 10447217
- [Background] Farber L, Stratz T, Bruckle W, Spath M, Pongratz D, Lautenschlager J, Kotter I, Zoller B, Peter HH, Neeck G, Alten R, Muller W. Efficacy and tolerability of tropisetron in primary fibromyalgia--a highly selective and competitive 5-HT3 receptor antagonist. German Fibromyalgia Study Group. Scand J Rheumatol Suppl. 2000;113:49-54. doi: 10.1080/030097400446643. PMID 11028832
- [Background] Spath M, Stratz T, Neeck G, Kotter I, Hammel B, Amberger CC, Haus U, Farber L, Pongratz D, Muller W. Efficacy and tolerability of intravenous tropisetron in the treatment of fibromyalgia. Scand J Rheumatol. 2004;33(4):267-70. doi: 10.1080/03009740410005818. PMID 15370724
- [Background] Ettlin T. Trigger point injection treatment with the 5-HT3 receptor antagonist tropisetron in patients with late whiplash-associated disorder. First results of a multiple case study. Scand J Rheumatol Suppl. 2004;119:49-50. PMID 15515414
- [Background] Muller W, Stratz T. Local treatment of tendinopathies and myofascial pain syndromes with the 5-HT3 receptor antagonist tropisetron. Scand J Rheumatol Suppl. 2004;119:44-8. PMID 15515413
- [Derived] Christidis N, Omrani S, Fredriksson L, Gjelset M, Louca S, Hedenberg-Magnusson B, Ernberg M. Repeated tender point injections of granisetron alleviate chronic myofascial pain--a randomized, controlled, double-blinded trial. J Headache Pain. 2015;16:104. doi: 10.1186/s10194-015-0588-3. Epub 2015 Dec 3. PMID 26634569